CLINICAL TRIAL: NCT05152680
Title: An Open-label, Single Dose, Mass Balance Study to Assess the Disposition of [14C]-NV-5138 in Healthy Male Subjects
Brief Title: Mass Balance Study of NV-5138 in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Navitor Pharmaceuticals, Inc. (Industry)
Collaborators: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAV-17A-006
Record Dates: First submitted 2021-11-03; First posted 2021-12-10 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-NV-5138 (Experimental): [14C]-NV-5138 oral solution
  Interventions: Drug: [14C]-NV-5138

INTERVENTIONS:
Drug: [14C]-NV-5138 — Single dose, given as oral solution, 1600 mg

SUMMARY:
The objective of this study is to assess the mass balance and routes of excretion of total radioactivity after a single oral dose of 1600 mg [14C]-NV-5138.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 40 to 65 years inclusive at the time of signing informed consent.
* Body mass index of 18.0 to 32.0 kg/m2 as measured at screening

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
* Subjects who are, or are immediate family members of, a study site or sponsor employee
* Evidence of current SARS-CoV-2 infection
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption of >21 units per week and (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Subjects with pregnant or lactating partners
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker shall participate in the study
* Subjects who have participated in an ADME study involving carbon-14 within 12 months of screening.
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are not allowed
* Clinically significant abnormalities on vital signs or ECGs as judged by the investigator at screening or pre-dose
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease or neurological disorder, as judged by the investigator
* Any history of major depression disorder (MDD) requiring treatment or counselling or any other clinically significant psychiatric history, as judged by the investigator
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) in the 14 days or 5 half-lives, whichever is longer, before IMP administration. COVID-19 vaccines are accepted concomitant medications. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
* Subject answers "yes" to "Suicidal Ideation" Items 1 or 2 on the C-SSRS at screening
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Cumulative total radioactivity in urine and faeces | urine and fecal samples up to 168 hours post dose
  The percentage of the radioactive dose recovered in urine, faeces and in total

SECONDARY OUTCOMES:
AUCinf for NV-5138, metabolite M8 and total radioactivity in plasma whole blood | up to 168 hours post-dose
  Area under the concentration-time curve from time zero (pre-dose) to infinity
AUClast for NV-5138, metabolite M8 and total radioactivity in plasma whole blood | up to 168 hours post-dose
  Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration
Cmax for NV-5138, metabolite M8 and total radioactivity in plasma whole blood | up to 168 hours post-dose
  Maximum observed concentration
Tmax for NV-5138, metabolite M8 and total radioactivity in plasma whole blood | up to 168 hours post-dose
  Time of maximum observed concentration
Tlast for NV-5138, metabolite M8 and total radioactivity in plasma whole blood | up to 168 hours post-dose
  Time of the last measurable concentration
t1/2 for NV-5138 and total radioactivity in plasma and whole blood | up to 168 hours post-dose
  Terminal elimination half-life
CL/F for NV-5138 in plasma | up to 168 hours post-dose
  Total oral clearance
Vz/F for NV-5138 in plasma | up to 168 hours post-dose
  Apparent volume of distribution
MPR Cmax in plasma | up to 168 hours post-dose
  metabolite to parent ration based on Cmax
MPR AUCinf in plasma | up to 168 hours post-dose
  metabolite to parent ration based on AUCinf
Whole blood to plasma partitioning for total radioactivity | up to 168 hours post-dose
  The AUCinf ratio of whole blood to plasma
CLR for NV-5138 | up to 168 hours post-dose
  Renal clearance
Ae for total radioactivity in urine and feces | up to 168 hours post-dose
  amount of total radioactivity excreted over each sampling period
%Dose for total radioactivity in urine and feces | up to 168 hours post-dose or until mass balance criteria have been met
  amount of total radioactivity eliminated in faeces expressed as a percentage of the radioactive dose administered over each sampling period
Incidence of treatment-emergent adverse events | through study completion at one week
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom